CLINICAL TRIAL: NCT02943772
Title: Effect of Local Cooling of Testis in Patient With Epididymitis on Analgetics Consumption and Pain Level
Brief Title: Does Local Cooling of Testis in Patients With Epididymitis Relieve Pain and Reduce Quantity of Analgetics Intake?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Dan Leibovici, professor, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0092-16-KMC
Record Dates: First submitted 2016-09-26; First posted 2016-10-25 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local hypothermia (Experimental): Local application of a brick cooled to -20(celsius)
  Interventions: Other: Local hypothermia
- Control (Sham Comparator): Local application of a brick in room temperature
  Interventions: Other: Control

INTERVENTIONS:
Other: Local hypothermia — Cooled brick
  Arms: Local hypothermia
Other: Control — Control brick
  Arms: Control

SUMMARY:
The investigators propose to examine the effect of local cooling of testis in participants with acute epididymitis or orchiepididymitis on participants reported pain level and analgetics consumption.

DETAILED DESCRIPTION:
Epididymitis or orchiepididymitis is an acute disease causing pain and discomfort.

our hypothesis is that local cooling of the affected testis or epididymis may relieve the pain and reduce the analgetics consumption In order to examine this hypothesis we will recruit adult patients with epididymitis or orchiepididymitis and will randomize these patients to two arms.

One arm will receive every 8 hours a brick cooled for at least 2 hours in -20(celsius) for local use on the affected hemiscrotum, while the second arm will receive a brick in room temperature.

Pain level will be estimated one hour following the application of the brick using visual analogue pain score. Patient will receive analgetics according to a predefined escalating protocol.

Pain level and analgetics consumption will be compared between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Male patients 18-99 years
* Acute epididymitis or acute orchiepididymitis

Exclusion Criteria:

* Patient unable to informed consent
* Suspicion of testicular malignancy

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-11-07 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
change in pain level | pain level change from baseline three times a day following the intervention of brick/cooled brick from randomization throughout the hospitalization for at least 24 hours of hospitalization and up to 50weeks
  intervention and measurement will be examined three times a day following brick/cooled brick

SECONDARY OUTCOMES:
Total consumption in grams of protocol analgetics | analgetics consumption will be recorded from randomization throughout the hospitalization for at least 24 hours of hospitalization and up to 50weeks
  each protocol Analgetic will be summarized individually in grams

CONTACTS AND LOCATIONS:
Overall Officials: Dan Leibovici, MD, Principal Investigator — Kapaln medical center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No